CLINICAL TRIAL: NCT05171140
Title: Influence of Different Spatial Distribution of Hollow Screws on Blood Supply and Prognosis of Femoral Neck Fractures in the Elderly
Brief Title: Influence of the Spatial Distribution of Hollow Screws on the Blood Supply and Prognosis of Femoral Neck Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020YJZX0112
Record Dates: First submitted 2021-11-22; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Femoral Neck Fracture
Keywords: Femoral Neck Fracture; Robot assisted; Blood supply of femoral head
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hollow nails are arranged in a triangle (Experimental): Hollow nails are arranged in a triangle
  Interventions: Procedure: Triangular Nail Placement of Femoral Neck
- Hollow nail inverted triangle arrangement (Experimental): Hollow nail inverted triangle arrangement
  Interventions: Procedure: Triangular Nail Placement of Femoral Neck

INTERVENTIONS:
Procedure: Triangular Nail Placement of Femoral Neck — Triangular Nail Placement of Femoral Neck in arm A Femoral Neck Inverted Triangle Nail Surgery in arm B

SUMMARY:
Femoral neck fracture is a common type of fracture in the elderly. For those without significant displacement (Garden I, II), more hip-preserving treatment strategies are adopted. The classic parallel hollow screw internal fixation for hip-preserving treatment is based on the sliding compression theory, and a clinical debate has gradually emerged, that is, the positive triangle And the two different spatial distribution methods of hollow nails and inverted triangle, which one is better. In addition, the distribution of hollow nails in actual operations is difficult to achieve a standard triangular distribution, and the damage to the epiphyseal vessels in the femoral head caused by repeated drilling of the guide needle cannot always be ignored. The relationship between the distribution and injury of blood vessels in the femoral head and the spatial distribution of hollow screws on the prognosis of head necrosis of non-displaced femoral neck fractures in the elderly is worth studying. This topic is based on the three advantages of TianJi orthopedic robots used in the elderly femoral neck fracture hollow nail hip-saving surgery: 1.standardized triangular nail placement with strong repeatability; 2. precise nail placement to reduce the risk of screw penetration; 3. limited guide pins The number of drill holes is to rule out repeated drill holes that damage the blood vessels in the femoral head. The preoperative and postoperative vascular injury in the femoral head (enhanced MRI of the femoral head) was compared to assess the prognosis of patients, and to clarify the influence of the spatial distribution of hollow screws on the blood supply and prognosis of the femoral neck fracture in the elderly.

DETAILED DESCRIPTION:
the investigators choose 60-80-year-old Garden I or II patients with initial fractures. Hollow nails are the first choice for treatment of these patients. However, the spatial arrangement of hollow nails, local blood supply, and biomechanical properties have a greater impact on the prognosis of fractures. , There are still some controversies, which are also the current research hotspots. Our research conclusions may increase the success rate of hip preservation and will guide the treatment of these patients. This study is based on the precise placement of nails by the Dimensity orthopedic robot, and compares the vascular injury of the femoral head before and after the nail placement (femoral head enhanced MRI) to assess the prognosis of the patient. The influence of blood supply and prognosis of femoral neck fracture in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* A new initial intracapsular fracture of the femoral neck;
* Garden classification I or II;
* Accept closed reduction robot-assisted hollow nail surgery;
* ASA score 1-2, can tolerate anesthesia;
* Age 60-80 years old (inclusive);
* Able to fully understand and voluntarily sign informed consent.

Exclusion Criteria:

* Old or pathological fractures;
* Patients with acetabular fracture;
* Those who have general conditions or accompanying diseases that make it difficult for people to tolerate surgery, such as: coagulation dysfunction, or heart, liver, and kidney dysfunction;
* Severe infections systemically or locally;
* Those who refuse to sign informed consent;
* In any case, if the researcher believes that the patient is not suitable for this treatment or there are other factors that affect the efficacy of the observation of this study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
comparison of hip joint function at 6 months | 6 months after surgery
  Harris score
comparison of hip joint function at 12 months | 12 months after surgery
  Harris score
Imaging evaluation of the vascular condition of the femoral head epiphysis before surgery | One day before surgery
  Imaging evaluation of the vascular condition of the femoral head epiphysis
Imaging evaluation of the vascular condition of the femoral head epiphysis after surgery | 2 months after surgery
  Imaging evaluation of the vascular condition of the femoral head epiphysis

SECONDARY OUTCOMES:
Intraoperative indicators-surgical blood loss | Intraoperative
  surgical blood loss（ml）
Intraoperative indicators-operation time | Intraoperative
  operation time（minute）

CONTACTS AND LOCATIONS:
Overall Officials: Ping Huang, Master, Principal Investigator — Shanghai Jiaotong University School of Medical Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No